CLINICAL TRIAL: NCT04292847
Title: LCCC1931: Interventions to Address Symptoms and Deficits in Women Age 70 Plus During the First Year Post Primary Treatment for Early Breast Cancer
Brief Title: LCCC1931:Post-treatment Intervention in Women With Breast Cancer (70y/o+)
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Breast Cancer Research Foundation (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: LCCC 1931; 5UG1CA233373-04 (NIH)
Record Dates: First submitted 2020-02-27; First posted 2020-03-03 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Geriatric Assessment: Participants fill out the geriatric assessment during a clinic visit and receive recommendations based on results
  Interventions: Other: Referrals Recommendations

INTERVENTIONS:
Other: Referrals Recommendations — All participants will complete the geriatric assessment and receive Referral recommendations based on the assessment.

SUMMARY:
This study recruits woman over the age of 70 who have completed primary treatment for early breast cancer in the last 2 months. A survey called the geriatric assessment will be used to identify symptoms and issues participants experience.This information will be given to the patient's medical oncology team, and used to make referrals to specialists. This study is designed to determine if these assessments and timely interventions can be completed during clinic visits, and determine if these participants comply with recommendations.

DETAILED DESCRIPTION:
1. Primary Objective Estimate the percent of patients with at least one deficit who agree to at least one referral. "Interest" in the intervention will be determined by this metric. This agreement will be determined within the 1-2 weeks of consenting to the study through interactions between patients and the Study Team.

This study will recruit 100 participants in 2 years. These participants will complete the geriatric assessment and be given recommendations based on results. The study team will follow the medical record to determine if the participants complied with the recommendations

ELIGIBILITY:
Inclusion Criteria:

* Women aged 70 or older
* within 6 months of complete primary treatment (surgery, chemotherapy, targeted therapy, or radiation) for breast cancer (Stage I-III)
* Able to read English
* Willing and capable of providing informed consent

Exclusion Criteria:

-Has dementia, altered mental status, or any psychiatric or co-morbid condition prohibiting the understanding or rendering of informed consent.

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Study Population: Patients are recruited within 6 months of completing primary treatment (surgery, chemotherapy, anti-HER-2 therapy, and/or radiation treatment).
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants who agree to referral | 3 years
  Number of participants who agree to suggested referral within 1-2 weeks of consent

SECONDARY OUTCOMES:
Percentage of referral acceptance among participants with function deficits, as identified by the geriatric assessment | 3 years
  Number of participants with function who agree to suggested referral within 1-2 weeks of consent compared to total number of participants with function deficits
Percentage of referral acceptance among participants with cognition deficits, as identified by the geriatric assessment | 3 years
  Number of participants with cognition who agree to suggested referral within 1-2 weeks of consent compared to total number of participants with cognition deficits
Percentage of referral acceptance among participants with mental health index deficits, as identified by the geriatric assessment | 3 years
  Number of participants with function mental health index who agree to suggested referral within 1-2 weeks of consent compared to total number of participants with mental health index deficits
Percentage of referral acceptance among participants with comorbidity deficits, as identified by the geriatric assessment | 3 year
  Number of participants with function comorbidity who agree to suggested referral within 1-2 weeks of consent compared to total number of participants with comorbidity deficits
Percentage of referral acceptance among participants with polypharmacy deficits, as identified by the geriatric assessment | 3 years
  Number of participants with function polypharmacy who agree to suggested referral within 1-2 weeks of consent compared to total number of participants with polypharmacy deficits
Percentage of referral acceptance among participants with Nutrition deficits, as identified by the geriatric assessment | 3 years
  Number of participants with function Nutrition who agree to suggested referral within 1-2 weeks of consent compared to total number of participants with Nutrition deficits

CONTACTS AND LOCATIONS:
Overall Officials: Hyman Muss, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials